CLINICAL TRIAL: NCT04182438
Title: Influence of Low Potassium Content Vegetables in End-Stage Renal Disease on Chronic Dialysis Patients
Brief Title: Low Potassium Content Vegetables in End-Stage Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsuan-Jen Lin, Nephrology physician doctor, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CMUH108-REC3-136
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: End-stage Renal Disease
Keywords: Low potassium content vegetables; End-Stage Renal Disease; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This study will enroll 40 End-Stage Renal Disease on chronic hemodialysis patients. We will perform a randomized, double-blind, cross over study. In one group, low potassium content vegetables use as study intervention for two weeks (study phase), then shift to placebo (ordinary vegetables) for two weeks. In another group, ordinary vegetables will use firstly, then change to low potassium content vegetable use. Serum potassium, blood pressure, and biochemistries will analyze at the end of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low potassium then normal potassium (Experimental): After giving the vegetables with low potassium content vegetables for 2 weeks, the serum potassium level was recorded; after 2 weeks of washing time, the normal potassium content vegetables was given for 2 weeks, and the serum potassium concentration was recorded and the test was terminated.
  Interventions: Dietary Supplement: Low potassium content vegetables
- Normal potassium then low potassium (Experimental): After giving the normal potassium content vegetables for 2 weeks, the serum potassium concentration was recorded; after 2 weeks of washing time, the low potassium content vegetables use for 2 weeks, then the serum potassium level was recorded at the time. The test was terminated.
  Interventions: Dietary Supplement: Low potassium content vegetables

INTERVENTIONS:
Dietary Supplement: Low potassium content vegetables — use low-potassium content vegetables

SUMMARY:
Hyperkalemia is common in End-Stage Renal Disease on chronic hemodialysis patients. The most common cause of mortality in End-Stage Renal Disease patients is sudden cardiac death caused by hyperkalemia. Hyperkalemia also increased urgent dialysis and hospitalization rate. Thus, the management for hyperkalemia in End-Stage Renal Disease patients is crucial, including restricting dietary potassium, medication control, and dialysis dosage adjustment. In the ordinary diet, the significant sources of potassium are vegetables and fruit. In our study, the investigators try to find out the influence of low potassium content vegetables for serum potassium control in End-Stage Renal Disease on chronic hemodialysis patients.

This study is a prospective cohort study; the investigators enroll forty End-Stage Renal Disease on hemodialysis patients and perform this study in eight weeks period. The investigators conduct a randomized, double-blind and cross-over trial for investigating the influence of low potassium content vegetables on End-Stage Renal Disease patients. The serum potassium level will record under different potassium content vegetables. The possible adverse effects of low potassium content vegetables, cardiac arrhythmia, will also obtain by chart records during this study.

DETAILED DESCRIPTION:
According to the plan moderator, after the patient agrees and signs the test consent form, the patients will be randomly divided into two groups. The screening execution time of this patient is expected to be 2 weeks. After randomization into two groups, the first group was given low potassium content vegetables for 2 weeks, and the serum potassium level was recorded during routine blood tests in the hemodialysis; then the normal potassium content vegetables was given after 2 weeks of washing time. After 2 weeks of normal potassium content vegetables, the serum potassium level was recorded during routine blood tests in the hemodialysis, and the test was terminated. The second group was given normal potassium content vegetables for 2 weeks, and the serum potassium level was recorded during routine blood tests in the hemodialysis; after 2 weeks of washing time, the low potassium content of the vegetables was given for 2 weeks. The serum potassium level was c, and the test was terminated. Compare the potassium concentration of blood in hemodialysis patients using low potassium vegetables with normal potassium content vegetables.

Routine blood test observed in this trial - including blood counts (white blood cells, red blood cells, platelet count, hemoglobin, hematocrit), blood biochemical tests (including urea nitrogen, creatinine, liver function, albumin, total protein, uric acid, electrolytes) (sodium, potassium, calcium, phosphorus, magnesium, iron), iron storage protein, fasting blood glucose, blood fat, parathyroid hormone concentration, dialysis parameters (artificial kidney, weekly dialysis times, dialysis hours, dialysate concentration, dialysis volume) , dialysate temperature), and the patient's blood pressure changes and arrhythmia occurred statistical analysis. Outpatient hemodialysis patients' medical records have been coordinated with the hospital electronic data, data obtained from electronic medical records to obtain patients with hypokalemia drugs or hypertension drug use records, dialysis records. All the information obtained will be linked to ensure patient privacy.

During the trial, if the patient has hospitalization for arrhythmia caused by hypokalemia, the record will be withdrawn from the trial and then withdrawn from the clinical trial and excluded from the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* End-Stage Renal Disease on chronic hemodialysis patients in single center

Exclusion Criteria:

* younger than 20 years old, the pregnant woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
Change of serum potassium level | two weeks
  Measure pre-dialysis serum potassium

CONTACTS AND LOCATIONS:
Locations (1):
- Asia University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No